CLINICAL TRIAL: NCT04893018
Title: Phase 1 Study of NT-I7 (rhIL-7-hyFc) for the Treatment of Kaposi Sarcoma in Patients With or Without Infection With HIV
Brief Title: NT-I7 for Kaposi Sarcoma in Patients With or Without HIV
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to end of funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Cancer Immunotherapy Trials Network (CITN) (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CITN-17; NCI-2021-01002 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UM1CA154967 (NIH)
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-04

CONDITIONS: AIDS-Related Kaposi Sarcoma; HIV Infection; Kaposi Sarcoma
MeSH Terms: conditions — AIDS-related Kaposi sarcoma; HIV Infections; Sarcoma, Kaposi | interventions — efineptakin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (efineptakin alfa) (Experimental): Patients receive efineptakin alfa IM on day 1. Cycles repeat every 9 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Efineptakin alfa

INTERVENTIONS:
Biological: Efineptakin alfa — Given IM
  Other Names: 2026634-47-7; GX-I7; Hyleukin-7 (TM); Il-7 Hybrid Fc; IL-7-hyFc; NT-I7; rhIL-7-hyFc

SUMMARY:
This phase I trial studies the best dose and effects of NT-I7 in treating Kaposi sarcoma in patients with or without HIV. NT-I7 works by using a patient's immune system to fight cancer. It is made in a laboratory and is used to boost, direct, or restore the body's natural defenses against cancer. NT-I7 may work better in treating Kaposi sarcoma.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study.

Patients receive efineptakin alfa intramuscularly (IM) on day 1. Cycles repeat every 9 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up on day 30 (+/- 7 days) and then every 12 weeks for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed Kaposi sarcoma
* Patients must have evaluable disease. Note: Kaposi sarcoma will be evaluated using a modified version (consistent with National Cancer Institute [NCI] studies) of the Acquired Immunodeficiency Syndrome (AIDS) Clinical Trial Group (ACTG) Oncology Committee staging and response definitions for KS
* No upper or lower limit on the number of prior therapies or stage of disease
* HIV-positive patients must have been on effective anti-retroviral (ART) therapy for at least 3 months prior to enrollment, with persistent KS affecting quality of life due to either T1 disease or T0 disease with inadequate disease regression on ART alone
* HIV-positive patients must have undetectable HIV viral loads =< 40 copies/mL measured using a Food and Drug Administration (FDA)-approved commercial assay with lower limit of detection between =< 20 copies/mL and =< 40 copies/mL
* Patients with visceral involvement must:

  * Meet other eligibility criteria
  * Have any/all associated tumor associated symptoms =< grade 2 by Common Terminology Criteria for Adverse Events (CTCAE) criteria; and/or
  * Require no immediate intervention (e.g. mild oozing of oral KS not an exclusion criteria)
* Patients must provide newly obtained core, punch, or excisional biopsy of a tumor lesion obtained up to 28 days prior to treatment initiation. An archival tumor sample obtained within 1 year of screening is allowed if pre treatment biopsy is deemed unsafe or technically not feasible
* Patients must be >= 18 years of age on day of signing informed consent document. Because no dosing or adverse event data are currently available on the use of NT-I7 in patients < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 2,500/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9/dL
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN) OR < 3 x institutional ULN for Gilbert's syndrome or HIV protease inhibitors
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional ULN
* Creatinine =< 2 x institutional ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 by Cockcroft-Gault. At the discretion of the treating physician, a 24-hour urine creatinine clearance could be obtained and utilized as the gold standard if creatinine clearance by Cockcroft-Gault is < 30 and prevents patient enrollment on the trial
* Patients with chronic hepatitis B virus (HBV) infection must be on suppressive antiviral therapy
* Patients with a history of hepatitis C virus (HCV) infection must have an undetectable HCV viral load due to prior treatment or natural resolution
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours before receiving the first dose of the study agent. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* The effects of NT-I7 on the developing human fetus are unknown. For this reason and because NT-I7 may have an adverse effect on pregnancy and poses risk to the human fetus, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 90 days after completion of NT-I7 administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy or other KS directed therapy other than ART for HIV within 2 weeks before the initiation of study treatment
* Patients who have not recovered from immune related adverse events due to prior therapy (i.e., have residual toxicities > grade 1) with the exception of hypothyroidism managed by supplemental levothyroxine
* Patients who have received treatment with any other investigational agent within 4 weeks before initiation of study treatment
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Patients who have a history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients who have received treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2, pomalidomide, or immune checkpoint inhibitors) within 6 weeks before initiation of study treatment
* Patients who have received treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor [anti-TNF] agents) within 2 weeks before initiation of study treatment

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled;
  * The use of inhaled corticosteroids, and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients who have a history or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis. Note: the following will NOT be exclusionary:

  * The presence of laboratory evidence of autoimmune disease (e.g., positive antinuclear antibody (ANA) titer or lupus anticoagulant) without associated symptoms
  * Clinical evidence of vitiligo or other forms of depigmenting illness
  * Mild autoimmunity not impacting the function of major organs (e.g., limited psoriasis)
* Patients with uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure (New York Heart Association Class III or IV), unstable angina pectoris, cardiac arrhythmia, recent myocardial infarction (within the last 6 months). Patients with known history of treatment with cardiotoxic agents, including anthracyclines, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification
* Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because the effects of NT-I7 on the developing human fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with NT-I7, breastfeeding should be discontinued if the mother is treated with NT-I7
* Patients with a history of solid organ or allogeneic stem cell transplant
* Patients with continuing KS regression on ART alone. Stable disease allowed
* Patients with a prior or concurrent malignancy requiring active therapy
* Patients with active tuberculosis
* Patients who have a history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening X-Ray. History of radiation pneumonitis in the radiation field (fibrosis) is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ching (Jackie) Wang, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramaswami R, Kask AS, D'Amico L, Menon MP, Lurain K, Yarchoan R, Ekwede I, Couey P, Burnham E, Angeldekao A, Ha Lee B, Kaiser JC, Cheever M, Uldrick TS, Kwok LL, Wright A, Fling SP, Wang CJ. Phase I study of efineptakin alfa (NT-I7) for the treatment of Kaposi sarcoma. J Immunother Cancer. 2025 Feb 6;13(2):e010291. doi: 10.1136/jitc-2024-010291. PMID 39915263

RESULTS

PARTICIPANT FLOW:
Groups:
- NT-I7 (Efineptakin Alfa) Dose Level 1: Participants receive 480 µg/kg NT-I7 (Efineptakin alfa) IM on day 1. Cycles repeat every 9 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  NT-I7 (Efineptakin alfa): Given IM
- NT-I7 (Efineptakin Alfa) Dose Level 2: Participants receive 960 µg/kg NT-I7 (Efineptakin alfa) IM on day 1. Cycles repeat every 9 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  NT-I7 (Efineptakin alfa): Given IM
Period: Overall Study
Arm/Group | NT-I7 (Efineptakin Alfa) Dose Level 1 | NT-I7 (Efineptakin Alfa) Dose Level 2
Started | 6 | 2
Completed | 2 | 0
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Study Terminated | 1 | 2

BASELINE CHARACTERISTICS:
Population: Population included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | NT-I7 (Efineptakin Alfa) Dose Level 1 | NT-I7 (Efineptakin Alfa) Dose Level 2 | Total
Number analyzed (Participants) | 6 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (7.2) | 37.0 (5.7) | 52.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: Measured by Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 30 days after last dose of NT-I7, approximately 31 weeks total
Population: Analysis is conducted on all enrolled participants who received at least one dose of NT-I7.
Measure: Number; unit: percentage of participants
Arm/Group | NT-I7 (Efineptakin Alfa) Dose Level 1 | NT-I7 (Efineptakin Alfa) Dose Level 2
Number analyzed (Participants) | 6 | 2
percentage of participants | 100 | 100

2. Secondary Outcome: Objective Response Rate (ORR).
Description: Defined as the proportion of participants who achieved Complete Response (CR) or Partial Response (PR) according to modified Acquired Immunodeficiency Syndrome (AIDS) Clinical Trials Group Criteria (ACTG) criteria.
Time Frame: 12 months
Population: Analysis is conducted on all enrolled participants who received at least one dose of NT-I7 and provided at least one post-baseline response assessment, and did not discontinue study treatment prior to the first protocol-specified timepoint for evaluation of response to therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | NT-I7 (Efineptakin Alfa) Dose Level 1 | NT-I7 (Efineptakin Alfa) Dose Level 2
Number analyzed (Participants) | 5 | 2
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 1 | 2
  Objective Response Rate (CR+PR) | 1 | 2

3. Secondary Outcome: Duration of Response (DOR)
Description: Measured in participants who obtain a partial response or better and defined as time from the best response within the first 36 weeks of therapy until disease progression or censoring. Kaplan Meier survival estimates constructed for each of these survival endpoints with 95% confidence intervals (CIs), for up to 1 year following initiation of treatment in all participants.
Time Frame: Up to 1 year
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NT-I7 (Efineptakin Alfa) Dose Level 1 | NT-I7 (Efineptakin Alfa) Dose Level 2
Number analyzed (Participants) | 5 | 2
months | NA [NA to NA] — Due to insufficient number of participants, median duration of response (DOR) could not be calculated, and upper and lower confidence interval for DOR could not be obtained using Kaplan-Meier estimates. | NA [NA to NA] — Due to insufficient number of participants, median duration of response (DOR) could not be calculated, and upper and lower confidence interval for DOR could not be obtained using Kaplan-Meier estimates.

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Defined as the time from administration of the first dose of NT-I7 until disease progression or death or censoring. Kaplan Meier survival estimates will be constructed for each of these survival endpoints with 95% CIs, for up to 1 year following initiation of treatment in all participants.
Time Frame: Assessed up to 1 year
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NT-I7 (Efineptakin Alfa) Dose Level 1 | NT-I7 (Efineptakin Alfa) Dose Level 2
Number analyzed (Participants) | 5 | 2
months | NA [2.1 to NA] — Due to insufficient number of participants, median progression free survival (PFS) could not be calculated. | NA [NA to NA] — Due to insufficient number of participants, median progression free survival (PFS) could not be calculated, and upper and lower confidence interval for PFS could not be obtained using Kaplan-Meier estimates.

5. Secondary Outcome: Overall Survival (OS)
Description: From administration of the first dose of NT-I7 until death or censoring. Kaplan Meier survival estimates will be constructed for each of these survival endpoints with 95% CIs.
Time Frame: Assessed up to 1 year following initiation of treatment
Population: Analysis is conducted on all enrolled and treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NT-I7 (Efineptakin Alfa) Dose Level 1 | NT-I7 (Efineptakin Alfa) Dose Level 2
Number analyzed (Participants) | 6 | 2
months | NA [NA to NA] — Due to insufficient number of participants, median overall survival (OS) could not be calculated, and upper and lower confidence interval for OS could not be obtained using Kaplan-Meier estimates. | NA [NA to NA] — Due to insufficient number of participants, median overall survival (OS) could not be calculated, and upper and lower confidence interval for OS could not be obtained using Kaplan-Meier estimates.

6. Secondary Outcome: Effect of NT-I7 on Kinetics of Absolute Lymphocyte Counts (ALC) in Blood
Description: For analysis of circulating lymphocytes, we will describe fold-change (median and range) in blood ALC. Fold change from baseline is defined as the ratio of the value at the visit to that at baseline.
Time Frame: From pre-administration to each time point following first administration (1, 4, and 9 weeks)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: No units, median and IQR of ratios
Arm/Group | NT-I7 (Efineptakin Alfa) Dose Level 1 | NT-I7 (Efineptakin Alfa) Dose Level 2
Number analyzed (Participants) | 5 | 2
No units, median and IQR of ratios
  Week 1 | 1.06 [0.62 to 1.10] | 1.15 [1.06 to 1.24]
  Week 4 | 3.20 [3.20 to 3.47] | 3.93 [3.29 to 4.58]
  Week 9 | 3.01 [2.65 to 3.12] | 3.24 [2.96 to 3.52]

7. Secondary Outcome: Effect of NT-I7 on Kinetics of CD4+ T Cells in Blood.
Description: Described by fold-change (median and range) in blood CD4+ T cells. Fold change from baseline is defined as the ratio of the value at the visit to that at baseline.
Time Frame: From pre-administration to each time point following first administration (1, 4, and 9 weeks)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: No units, median and IQR of ratios
Arm/Group | NT-I7 (Efineptakin Alfa) Dose Level 1 | NT-I7 (Efineptakin Alfa) Dose Level 2
Number analyzed (Participants) | 4 | 2
No units, median and IQR of ratios
  Week 1 | 1.26 [0.76 to 1.71] | 1.19 [0.84 to 1.54]
  Week 4 | 4.46 [3.07 to 5.92] | 6.30 [4.95 to 7.66]
  Week 9 | 3.26 [2.18 to 4.19] | 4.45 [3.42 to 5.47]

8. Secondary Outcome: Effect of NT-I7 on Kinetics of CD8+ T Cells in Blood.
Description: Described by fold-change (median and range) in blood CD8+ T cells. Fold change from baseline is defined as the ratio of the value at the visit to that at baseline.
Time Frame: From pre-administration to each time point following first administration (1, 4, and 9 weeks)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: No units, median and IQR of ratios
Arm/Group | NT-I7 (Efineptakin Alfa) Dose Level 1 | NT-I7 (Efineptakin Alfa) Dose Level 2
Number analyzed (Participants) | 4 | 2
No units, median and IQR of ratios
  Week 1 | 0.89 [0.78 to 1.14] | 1.29 [1.27 to 1.32]
  Week 4 | 3.25 [2.43 to 4.48] | 4.12 [3.45 to 4.79]
  Week 9 | 2.53 [1.84 to 3.42] | 3.28 [2.93 to 3.64]

9. Other Pre Specified Outcome: Immunogenicity of NT-I7
Description: The proportion of participants developing neutralizing antibodies will be summarized.
Time Frame: Up to 12 months after last dose of NT-I7
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed through study completion, up to 12 months; serious adverse events and other (not including serious) adverse events were assessed from the time of the first dose until 30 days after the last dose of NT-I7, approximately 31 weeks total.
Arm/Group | NT-I7 (Efineptakin Alfa) Dose Level 1 | NT-I7 (Efineptakin Alfa) Dose Level 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/2
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NT-I7 (Efineptakin Alfa) Dose Level 1 (N=6) | NT-I7 (Efineptakin Alfa) Dose Level 2 (N=2)
Injection site reaction (General disorders) | 1 | 0 — Administration site condition
Bacteremia (Infections and infestations) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NT-I7 (Efineptakin Alfa) Dose Level 1 (N=6) | NT-I7 (Efineptakin Alfa) Dose Level 2 (N=2)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Axillary lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Anal pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 1 | 1
Flu like symptoms (General disorders) | 0 | 1
Generalized edema (General disorders) | 0 | 1
Injection site reaction (General disorders) | 4 | 1
Localized edema (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 1
Herpes simplex reactivation (Infections and infestations) | 1 | 0
Papulopustular rash (Infections and infestations) | 1 | 0
Prostate infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 1
CD4 Lymphocytes decreased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 0
Lymphocyte count increased (Investigations) | 3 | 1
Neutrophil count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 2 | 0
Thyroid stimulating hormone increased (Investigations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Genital edema (Reproductive system and breast disorders) | 0 | 1
Right breast enlargement (Reproductive system and breast disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Flushing (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Enrollment for this study was terminated early due end of funding. Some of the planned statistical analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04893018/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT04893018/ICF_000.pdf